CLINICAL TRIAL: NCT02099747
Title: A Prospective Randomized Multicenter Study Comparing Horse Antithymocyte Globuline (hATG) + Cyclosporine A (CsA) With or Without Eltrombopag as Front-line Therapy for Severe Aplastic Anemia Patients.
Brief Title: hATG+CsA vs hATG+CsA+Eltrombopag for SAA
Acronym: RACE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: Novartis (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EBMT-RACE; 2014-000363-40 (EudraCT Number)
Record Dates: First submitted 2014-03-06; First posted 2014-03-31 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Severe Aplastic Anemia
Keywords: Aplastic Anaemia; Eltrombopag; HATG; ATGAM
MeSH Terms: conditions — Anemia, Aplastic | interventions — Antilymphocyte Serum; eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hATG + CsA (Active Comparator): Control Arm
  Interventions: Drug: hATG; Drug: CsA
- hATG + CsA + Eltrombopag (Experimental): Experimental
  Interventions: Drug: hATG; Drug: CsA; Drug: Eltrombopag

INTERVENTIONS:
Drug: hATG
  Other Names: ATGAM
Drug: CsA
Drug: Eltrombopag
  Arms: hATG + CsA + Eltrombopag

SUMMARY:
The null hypothesis of no difference in CR% at 3 months between the arms will be tested against the alternative of a difference in CR% at an alpha level of .05 by assessing the odds ratio for arm yielded by this model.

DETAILED DESCRIPTION:
This is a superiority trial aiming to increase the 3 month complete response rate. The sample size is calculated on the hypothesis that the experimental treatment will increase the 3 months response rate up to 21% (by 3 folds, based on the 7% reported in Scheinberg et al [17]). Under these assumptions, the sample size to reject the null hypothesis is n=96 patients for each treatment arm, increased by 4% for possibly not evaluable patients (total number of 200 patients, 100 each treatment arm). Statistical design for sample size calculation: increase from 7% (control arm) to 21% (investigational arm) in 3 month complete response rate (two-sided binomial test); alpha-error 0.05; power 0.8.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of severe or very severe aplastic anemia, defined by [29]:

   * At least two of the following:

     * Absolute neutrophil counts <0.5 x 109/L (severe) or <0.2 x 109/L (very severe)
     * Platelet counts <20 x 109/L
     * Reticulocyte counts <60 x 109/L
   * Hypocellular bone marrow (<30% cellularity), without evidences of fibrosis or malignant cells
2. Male or female age > 14 years;
3. Written informed consent
4. Willing and able to comply with all of the requirements and visits in the protocol
5. Understands that they can be randomised to either treatment arm
6. Negative pregnancy test for women of child bearing age
7. Written acceptance to use contraception (hormonal or barrier method of birth control; abstinence) for the entire duration of study participation.

Exclusion Criteria:

1. Prior immunosuppressive therapy with ATG (horse of rabbit) or any other lymphocyte depleting agent (i.e., alemtuzumab)
2. Eligibility to a sibling allogeneic stem cell transplantation
3. Evidence of a myelodysplastic syndrome, defined by the presence of myelodysplastic features, excess of blasts or karyotypic abnormalities typical of MDS (according to revised WHO 2008 criteria) [30],, as well as other primitive marrow disease. Patients with diagnosis of AA with cytogenetic abnormalities which are recurrent in MDS (according to revised WHO 2008 criteria) [30] should be included in this category, and are not eligible for the study; patients with del(20q), +8 and -Y are not included in this category, and thus are eligible for this study. The list of karyotypic abnormalities which qualifies for the diagnosis of MDS are listed in the Appendix.
4. History or clinical suspect of constitutional aplastic anemia (i.e. Fanconi Anemia with positive DEB/MMC test or Dyskeratosis Congenita)
5. History of malignant tumors with active disease within 5 years from enrollment, and/or previous chemo-radiotherapy
6. Previous history of stem cell transplantation
7. Treatment with cyclosporin A unless

   * <4 weeks of cyclosporin A treatment before enrolement and
   * wash out period of 2 weeks before enrollment
8. CMV viremia, as defined by positive PCR or pp65 test
9. WHO performance status ≥3
10. Pregnant or breast feeding patients
11. Patients with hepatic, renal or cardiac failure, or any other life- threatening concurrent disease
12. Patients with HIV infection
13. Patients without social health care assistance
14. Participation in another clinical trial within 1 month before the start of this trial
15. Patients and/or female partners of male patients not using highly effective method of birth control i.e. intrauterine device (IUD), hormonal (oral pill, injection, implants), tubal ligation or partner's vasectomy
16. subjects with known hypersensitivity to any of the component medications

The presence of a Paroxysmal Nocturnal Hemoglobinuria clone is not an exclusion criterion.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
CR rate | 3 months
  The primary objective of this trial is to investigate whether Eltrombopag added to standard immunosuppressive treatment increases the rate of early (at three months) complete response in untreated AA patient.

SECONDARY OUTCOMES:
Time to best heamatological response | 2 year
Heamatological Response at 6, 12, 18 and 24 months | 2 year
Cumulative incidence of response | 2 year
Overall survival | 2 year
Event-free survival | 2 year
Cumulative incidence of relapse rate | 2 year
Cumulative incidences of clonal evolution | 2 year
Cumulative incidence of PNH population occurrence and clinical hemolytic PNH occurrence | 2 year
Cumulative incidence of discontinuation of immunosuppressive therapy | 2 year
Rate of CsA-independent hematological response at 24 months | 2 year
Need for transfusions and number of transfusions required from treatment | 2 year
Need for any supportive care | 2 year
Comparison of number of SAEs between the two arms | 2 year
  To look for the safety and tolerability of the investigational treatment

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Risitano, MD, PhD, Principal Investigator — Federico II Medical School, Haematology Division, Napels; Regis Peffault de Latour, MD, PhD, Principal Investigator — St. Louis Hospital, Haematology Division, Paris
Locations (29):
- France (7):
  - Hopital Jean Minjoz, Besançon
  - Hôpital Haut-Lévèque, Bordeaux
  - Hôpital Huriez, Lille
  - Centre Hospitalier Lyon-Sud, Lyon
  - St. Louis Hospital, Paris
  - Pontchaillou Hospital, Rennes
  - Hôpital Purpan, Toulouse
- Italy (7):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Istituto G. Gaslini children's Hospital, Genova
  - San Martino Hospital, Genova
  - Fondazione IRCCS ca Granda Ospedale, Milan
  - 'Federico II' Medical School, Naples
  - La Sapienza University Hospital, Rome
  - AOU Città della Salute e della Scienza di Torino, Turin
- Netherlands (4):
  - AMC, Amsterdam
  - UMCG, Groningen
  - Leiden University Medical Center, Leiden
  - UMCU, Utrecht
- Spain (4):
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Institut Català d'Oncologia - Hospital Duran i Reynals, Barcelona
  - Donostia Hospital, Donostia / San Sebastian
  - Hospital La Fe, Valencia
- Switzerland (3):
  - University Hospital Basel, Basel
  - University Hospital Bern, Bern
  - University Hospital Zürich, Zurich
- United Kingdom (4):
  - St. James Hospital, Leeds
  - King's College Hospital, London
  - St. Bartholomew's Hospital, London
  - City Hospital, Nottingham

REFERENCES:
- [Derived] de Latour RP, Kulasekararaj A, Iacobelli S, Griffin M, Halkes CJ, Dufour C, Risitano AM. Plain language summary of RACE study results: addition of eltrombopag to standard treatment of severe aplastic anemia. Immunotherapy. 2024 Feb;16(3):135-142. doi: 10.2217/imt-2023-0200. Epub 2023 Dec 13. PMID 38088156
- [Derived] Peffault de Latour R, Kulasekararaj A, Iacobelli S, Terwel SR, Cook R, Griffin M, Halkes CJM, Recher C, Barraco F, Forcade E, Vallejo JC, Drexler B, Mear JB, Smith AE, Angelucci E, Raymakers RAP, de Groot MR, Daguindau E, Nur E, Barcellini W, Russell NH, Terriou L, Iori AP, La Rocca U, Sureda A, Sanchez-Ortega I, Xicoy B, Jarque I, Cavenagh J, Sicre de Fontbrune F, Marotta S, Munir T, Tjon JML, Tavitian S, Praire A, Clement L, Rabian F, Marano L, Hill A, Palmisani E, Muus P, Cacace F, Frieri C, van Lint MT, Passweg JR, Marsh JCW, Socie G, Mufti GJ, Dufour C, Risitano AM; Severe Aplastic Anemia Working Party of the European Society for Blood and Marrow Transplantation. Eltrombopag Added to Immunosuppression in Severe Aplastic Anemia. N Engl J Med. 2022 Jan 6;386(1):11-23. doi: 10.1056/NEJMoa2109965. PMID 34986284